CLINICAL TRIAL: NCT03252158
Title: Impact of the Availability of Healthier vs. Less Healthy Foods and Beverages on Purchasing From Hospital Vending Machines
Brief Title: Altering the Availability of Healthier vs. Less Healthy Items in Vending Machines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cambridge (Other)
Collaborators: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Rachel Pechey, Senior Research Associate, University of Cambridge
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PRE.2017.029
Record Dates: First submitted 2017-08-09; First posted 2017-08-17 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Healthy Diet

STUDY DESIGN:
Intervention Model Description: An adapted multiple treatment reversal design will be used, in which the number of slots containing (i) less healthy items and (ii) healthier items are altered over eight 4-week periods.
  Vending machines will be randomly allocated to one of two groups: (1) decreasing less healthy foods first or (2) decreasing healthier foods first.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decrease less healthy item availability (Experimental): Intervention: Availability of healthier vs. less healthy foods
  Remove less healthy items in 20% of slots, then fill the empty slots with healthier items.
  Interventions: Behavioral: Availability of healthier vs. less healthy foods
- Decrease healthier item availability (Experimental): Intervention: Availability of healthier vs. less healthy foods
  Remove healthier items in 20% of slots, then fill the empty slots with less healthy items.
  Interventions: Behavioral: Availability of healthier vs. less healthy foods

INTERVENTIONS:
Behavioral: Availability of healthier vs. less healthy foods — Altering the number of slots containing (a) healthier and (b) less healthy foods or beverages in hospital vending machines.
  Changes follow a 2-step process whereby decreases are implemented in a separate study period prior to increases in the contrasting group. Following a 4-week baseline period, all vending machines will be standardised to have 75% healthier drinks and/or 25% healthier snacks (study period 1). Vending machines will be randomly allocated to the order in which they: (1) decrease less healthy foods and increase healthier foods or (2) decrease healthier foods and increase less healthy foods (study periods 2&3 and 5&6). After each decrease-increase pair, machines will return to the standardised 75% healthier drinks / 25% healthier snacks (study periods 4 and 7).

SUMMARY:
Background: While there is some evidence that increasing the range of healthier foods and drinks and/or decreasing the range of less healthy options may increase healthier choices, more work is needed to establish the reproducibility of any effect. The current study aims to investigate the impact of altering the availability of healthier and less healthy foods and cold beverages in hospital vending machines.

Methods: An adapted multiple treatment reversal design will be used, in which all standard vending machines serving snack foods and/or cold beverages in one hospital in England change the number of slots containing (i) less healthy items and (ii) healthier items over eight 4-week periods. Changes will take place in a two-step process whereby decreases are implemented in a separate study period prior to increases in the contrasting food group. Following a 4-week baseline period, all vending machines will be standardised to have 75% healthier drinks and/or 25% healthier snacks (study period 1). Vending machines (n=9) will be randomly allocated to the order in which they: (1) decrease less healthy foods and increase healthier foods or (2) decrease healthier foods and increase less healthy foods (study periods 2&3 and 5&6). After each decrease-increase pair, machines will return to the standardised 75% healthier drinks and 25% healthier snacks (study periods 4 and 7). Sales data will be obtained via records of machine restocking.

Planned Analysis: The impact of the availability intervention will be assessed in separate linear mixed models for cold drinks and snacks, examining the impact on total energy (kcal) purchased, per restocking interval, with random effects for vending machine.

ELIGIBILITY:
Inclusion Criteria:

* All vending machines at one UK hospital selling standard-fare (i.e. not healthier alternatives) cold beverages and snack foods

Exclusion Criteria:

* Healthier alternative vending machines; vending machines selling hot drinks or meals

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-08-17 (Actual); Primary Completion 2018-03-28 (Actual); Study Completion 2018-03-28 (Actual)

PRIMARY OUTCOMES:
Energy purchased | Restocking interval (between 2-4 days; restocking occurs on set weekdays for each machine, to match usual restocking)
  Energy purchased (kcal) per restocking interval from intervention (standard-fare) vending machines

SECONDARY OUTCOMES:
Number of items sold | Restocking interval (between 2-4 days; restocking occurs on set weekdays for each machine, to match usual restocking)
  Number of items sold per restocking interval from intervention (standard-fare) vending machines
Energy purchased (healthier alternative machines) | Restocking interval (between 2-4 days; restocking occurs on set weekdays for each machine, to match usual restocking)
  Energy purchased (kcal) per restocking interval from non-intervention (healthier-fare) vending machines
Number of items sold (healthier alternative machines) | Restocking interval (between 2-4 days; restocking occurs on set weekdays for each machine, to match usual restocking)
  Number of items sold per restocking interval from non-intervention (healthier-fare) vending machines

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Pechey, PhD, Principal Investigator — University of Cambridge
Locations (1):
- University of Cambridge, Cambridge, Cambridgeshire, United Kingdom